CLINICAL TRIAL: NCT06084507
Title: Food Effects Study of GST-HG171 Tablets Combined With Ritonavir in Healthy Chinese Participants
Brief Title: Food Effects of GST-HG171 Tablets Combined With Ritonavir in Healthy Chinese Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fujian Akeylink Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GST-HG171-I-06
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Respiratory Infection
MeSH Terms: interventions — Ritonavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Single oral dose of ritonavir at -12 hours prior to GST-HG171/ritonavir dosing, followed by single oral dose of GST-HG171/ritonavir under fasted conditions. Ritonavir will continue to be dosed at 12 hours and 24 hours GST-HG171 dosing.
  Interventions: Drug: GST-HG171/ritonavir; Drug: ritonavir
- Treatment B (Experimental): Single oral dose of ritonavir at -12 hours prior to GST-HG171/ritonavir dosing, followed by single oral dose of GST-HG171/ritonavir under fed conditions. Ritonavir will continue to be dosed at 12 hours and 24 hours GST-HG171 dosing.
  Interventions: Drug: GST-HG171/ritonavir; Drug: ritonavir

INTERVENTIONS:
Drug: GST-HG171/ritonavir — Single oral dose of GST-HG171 300 mg (2 × 150 mg tablets)/ritonavir 100 mg under fed or fasted conditions at 0 hour on Day 1
Drug: ritonavir — Single oral dose of ritonavir 100 mg at -12 hours prior to GST-HG171/ritonavir dosing, and ritonavir 100 mg will be dosed at 12 hours and 24 hours after GST-HG171/ritonavir dosing.

SUMMARY:
A single-center, randomized, open, single-dose, two-cycle, two-sequence, cross-over study was conducted to evaluate the effect of food on the pharmacokinetic characteristics of GST-HG171 in combination with Ritonavir.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial and fully understand the content, process and possible adverse reactions of the trial;
2. Ability to complete research in accordance with test plan requirements;
3. Subjects (including partners) are willing to take effective pregnancy avoidance measures within 6 months after screening to the last study drug administration;
4. Male and female healthy subjects aged 18 to 50 years (including 18 and 50 years old);
5. Male subjects weigh no less than 50 kg, and female subjects weigh no less than 45 kg. Body mass index (BMI) = body weight (kg) / height 2 (m2), body mass index is in the range of 18 ~ 28 kg / m2 (including critical value);
6. Physical examination, normal or abnormal vital signs have no clinical significance

Exclusion Criteria:

1. Allergies (multiple drugs and food allergies);
2. Those who smoked more than 5 cigarettes per day in the 3 months before the trial;
3. Have a history of drug abuse and / or alcoholism (drink 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
4. Blood donation or massive blood loss (> 400 mL) within three months before screening;
5. Have a history of dysphagia or any gastrointestinal disease that affects drug absorption, including a history of frequent nausea or vomiting caused by any cause;
6. Have any disease that increases the risk of bleeding, such as hemorrhoids, acute gastritis, or gastric and duodenal ulcers;
7. Have taken the study drug or participated in the drug clinical trial within three months before taking the study drug;
8. Have Intended to take any drug that changes the activity of drug metabolizing enzyme 28 days before screening or during the study, including strong inhibitors and inducers that affect the metabolizing enzyme;
9. Took any prescription drugs or herbs within 14 days before screening, or took over-the-counter drugs or any vitamin products within 7 days before screening;
10. Vaccinated within 14 days before screening or planned to be vaccinated during the study;
11. Those who have taken special diets (including dragon fruit, mango, grapefruit, etc.) or have vigorous exercise or other factors affecting drug absorption, distribution, metabolism, excretion, etc. within 2 weeks before screening;
12. Those who cannot tolerate high fat (about 50% of the total calories) and high calorie (about 800~1000 calories) standard meals (only applies to subjects participating in the food effect study);
13. Abnormal ECG has clinical significance;
14. Female subjects were breastfeeding or had a positive serum pregnancy result during the screening period or during the study;
15. Clinical laboratory examinations are abnormal and clinically significant, or find the following diseases with clinical significance (including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, Immune, mental or cardiovascular disease) within 6 months before screening;
16. Positive screening for viral hepatitis (including hepatitis B and C), AIDS antigen / antibody, and Treponema pallidum antibody;
17. Acute disease or concomitant medication occurs from the screening stage to before study medication;
18. Ingested chocolate, any caffeinated or xanthine-rich food or drink 24 hours before taking the study drug;
19. People who have a positive urine drug screen or have a history of drug abuse or have used drugs within the past five years;
20. The investigator believes that there are other subjects who are not suitable for participating in this trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-12-27 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day 1 pre-dose, 0.25、0.5、0.75、1、1.25、1.5、2、3、4、6、8、12、24、48 and 72 hour post-dose
  Maximum Observed Plasma Concentration (Cmax) of GST-HG171
AUCinf | Day 1 pre-dose, 0.25、0.5、0.75、1、1.25、1.5、2、3、4、6、8、12、24、48 and 72 hour post-dose
  Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of GST-HG171
AUClast | Day 1 pre-dose, 0.25、0.5、0.75、1、1.25、1.5、2、3、4、6、8、12、24、48 and 72 hour post-dose
  Area Under the Curve From Time Zero o Last quantifiable concentration (AUClast) of GST-HG171

SECONDARY OUTCOMES:
urine | 120 hours from GST-HG171 administration
  Total recovery of GST-HG171 -related substances in urine
feces | 120 hours from GST-HG171 administration
  Total recovery of GST-HG171 -related substances in feces

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No